CLINICAL TRIAL: NCT06998277
Title: Impact of the Novel UC-TREAT Diet on the Gut Microbiome and Its Acceptability in Healthy Adults and Adults With Quiescent Ulcerative Colitis
Acronym: UC-TREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Professor, University of Glasgow
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-TREAT
Record Dates: First submitted 2025-05-09; First posted 2025-05-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; Dietary therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Two groups of participants. Adults with ulcerative colitis and healthy adult volunteers; both groups receive the same dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adults with quiescent Ulcerative Colitis (Experimental): Adults with Ulcerative Colitis currently in remission (SCCAI ≤ 5)
  Interventions: Other: Dietary therapy
- Healthy controls (Experimental): Healthy adults (≥ 16y)
  Interventions: Other: Dietary therapy

INTERVENTIONS:
Other: Dietary therapy — Participants with quiescent UC will undergo a 10-day "observational" period followed by 15-days of the UC-TREAT dietary intervention. Disease activity, quality of life, and gastrointestinal symptoms will be assessed throughout
  Arms: Adults with quiescent Ulcerative Colitis
Other: Dietary therapy — Healthy participants will undergo a 10-day "observational" period, followed by 15-days of the UC-TREAT dietary intervention. Gastrointestinal symptoms will be assessed throughout.
  Arms: Healthy controls

SUMMARY:
This will be an open-label dietary intervention study recruiting both healthy adults (≥16y) and adults with quiescent Ulcerative Colitis (UC). The study will span a total of 25 days and is divided into two phases; a 10-day run-in observation period (day -10 to day 0), during which the participant continues with their normal diet, and a 15-day dietary intervention period (day 0 to day 15), during which they will consume a diet high in specific high-fibre foods, fermented foods, berries, and a multivitamin-multimineral tablet. Throughout the study, participants will be asked to provide 3 blood samples (at days -10, 0, and 15), 4 stool and urine samples (at days -15, 0, 10, and 15), and to record a total of 6 days of food intake in provided food diaries. Disease activity, gastrointestinal symptoms, and quality of life will be assessed on 4 occasions (days -10, 0, 10, and 15) via validated questionnaires, and diet acceptability will be assessed at the end of the study.

DETAILED DESCRIPTION:
This will be an open-label dietary intervention study recruiting both healthy adults (≥16y) and adults with quiescent Ulcerative Colitis (UC) . The study will span a total of 25 days and is divided into two phases; a 10-day "run-in" observational period and a 15-day dietary intervention period.

During the 10-day "run-in" observational period (day -15 to day 0), participants will be asked to continue with their regular habitual diet and record their food intake in a provided estimated weight food diary with food photography for the first 3 of the 10 days. After this "run-in" period, participants will start the 15-day UC-TREAT dietary intervention (day 0 to day 15), where they will consume daily micronutrient supplements, increase intake of berries, and gradually increase intake of dietary fibre and fermented foods.

For the first 5 days of the dietary intervention, participants will enter a "ramping" phase, where, with the guidance of the researchers, they will consume 2 portions of berries (blueberries and raspberries) and 1 multivitamin-multimineral tablet each day. Participants will increase their fibre intake by 1 serving of high-fibre food per day until they reach an additional intake of 35g/d and increase fermented food intake by approximately 1 serving per day until they reach at least 5 servings per day. For the final 10 days of the UC-TREAT dietary intervention, participants will enter a "maintenance phase", where they will maintain this additional 35g of fibre intake and at least 5 servings of fermented foods daily. Participants will be asked to record 3 days of food intake in the provided food diaries during this period. The purpose of the ramping period is to reduce the sudden onset of functional abdominal symptoms typically associated with a rapid increase in dietary fibre consumption, including flatulence, bloating, and abdominal cramping. Throughout the study, participants will be asked to provide 3 blood samples (at days -10, 0 and 15), 4 stool and urine samples (at days -10, 0, 10, and 15), and to record a total of 6 days of food intake in provided food diaries.

On 4 occasions (days -10, 0, 10, and 15), all participants will be asked to complete a questionnaire assessing their gastrointestinal symptoms (GSRS-IBS), while participants with UC will also be asked to complete a questionnaire assessing their disease-specific quality of life (sIBDQ) and self-reported disease activity (SCCAI). At the end of the study (day 15), all participants will also be asked to complete an acceptability questionnaire to assess their tolerance of the diet.

ELIGIBILITY:
Inclusion Criteria:

Individuals with Ulcerative Colitis:

* Confirmed diagnosis of Ulcerative Colitis
* ≥16 years of age
* Motivated to follow the prescribed diet for the study period

Healthy controls:

* ≥16 years of age
* Motivated to follow the prescribed diet for the study period

Exclusion Criteria:

Individuals with Ulcerative Colitis:

* Self-reported active disease (SCCAI≥5) and/or a score ≥2 on any variable within SCCAI
* Previous surgery related to their UC (e.g. colectomy)
* Adjustment of medication dose in the previous month
* Initiation of a new medication in the prior 3 months
* BMI≥35kg/m2
* Pregnancy or lactation
* Regular use of pre/probiotic supplements
* Antibiotics or steroid use in the past 2 months
* Weight fluctuations ≥ 2kg in the past month
* Dietary restrictions (vegetarian, vegan, gluten-free etc)
* Participation in other interventional research.

Healthy controls:

* Regular use of medication or regular visits to a physician
* History of gut surgery
* BMI≥35kg/m2
* Pregnancy or lactation
* Regular use of pre/probiotic supplements
* Antibiotics or steroid use in the past 2 months
* Weight fluctuations ≥ 2kg in the past month
* Dietary restrictions (vegetarian, vegan, gluten-free etc)
* Participation in other interventional research.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in faecal butyrate concentration | At day -10, day 0, day 10, and day 15
  Change faecal butyrate concentration at the end of the diet (day 15) compared to baseline (day 0) and control (day -10).
Gastrointestinal symptoms | At day -10, day 0, day 10, and day 15
  Change in gastrointestinal symptoms compared to baseline, assessed via the GI Symptom Rating Scale (GSRS-IBS), will be used to assess GI tolerance of the diet. The GSRS-IBS assesses GI symptoms in 5 domains: pain, bloating, constipation, diarrhoea, and satiety, where a score increase indicates symptom increase.

SECONDARY OUTCOMES:
Faecal metabolites | At day -10, day 0, day 10, and day 15.
  Targeted faecal metabolites will be assessed via gas chromatography, colorimetry, and NMR metabolomics to evaluate changes to the faecal metabolome throughout the study period
Faecal microbiota diversity | At day -10, day 0, day 10, and day 15
  Change in faecal microbiota alpha-diversity during the diet compared to baseline and control.
Faecal microbiota composition | At day -10, day 0, day 10, and day 15
  Change in faecal microbiota composition (beta-diversity and taxa abundance) during the diet compared to baseline and control, as well as the differences between participants with UC and healthy controls.
Faecal calprotectin | At day -10, day 0, day 10, and day 15.
  Faecal calprotectin will be measured in all participants to assess any changes in gut inflammation throughout the study.
Blood inflammatory markers | At day -10, day 0 and day 15.
  Biomarkers of inflammation in plasma, such as C-reactive protein, will be measured in fasted blood samples.
Clinical disease activity | At day -10, day 0, day 10, and day 15.
  Clinical disease activity will be assessed via the Simple Clinical Colitis Activity Index (SCCAI), where a score increase indicates disease worsening and a score ≥ 5 indicates active disease.
Diet acceptability | Once at the end of the study period (day 15).
  Acceptability of the diet will be assessed in all participants at the end of the study, using a study specific 9-item questionnaire employing a 5-point likhert scale ("Strongly Agree", "Agree", "No opinion", "Disagree", "Strongly Disagree").
Quality of life (sIBDQ) | At day -10, day 0, day 10, and day 15.
  Quality of life will be assessed in participants with Ulcerative Colitis via the short-Inflammatory Bowel Disease Questionnaire (sIBDQ). This questionnaire assesses QoL in 4 domains: bowel, social, emotional, and systemic, where a score increase indicates improve quality of life.
Dietary adherence | Throughout the dietary intervention period (~15 days).
  Adherence to the prescribed diet will be assessed using daily food checklists.
Dietary intake | 3 days on 2 occasions (6 days in total) throughout the entire study period (~25 days).
  Dietary intake will be assessed via 3-day, estimated-portion food diaries supplemented with food photography. Food diaries will be recorded during the observational phase and during the dietary intervention phase of the study.
Stool form | At day -10, day 0, day 10, and day 15.
  Bristol Stool Chart Rating (BSCR) and percentage water content will be assessed to inform of any changes to stool form throughout the study.
Body composition | At day -10, day 0 and day 15.
  BMI and %fat mass will be assessed throughout the study to evaluate any changes to body composition throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gerasimidis, Principal Investigator — University of Glasgow; Athanasios Koutsos, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided